CLINICAL TRIAL: NCT06980129
Title: RITH4Hips - Rehabilitation in the Home After Hip Fracture
Brief Title: Rehabilitation in the Home After Hip Fracture
Acronym: RITH4Hips
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South West Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Thuy Anh Bui, Principal Investigator, South West Sydney Local Health District
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2025_ETH00123; 2025_ETH00123 (Other: South West Sydney Local Health District)
Record Dates: First submitted 2025-04-13; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Hip Fractures (ICD-10 72.01-72.2); Rehabilitation Program
Keywords: rehabilitation program; hip fracture
MeSH Terms: conditions — Hip Fractures | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: This study is a pragmatic, multicentre, randomised, single-blinded, two-group parallel, non-inferiority trial with an embedded qualitative component. Participants will be recruited in parallel from two different hospitals, ensuring a diverse and representative sample.
Who Masked: Outcomes Assessor
Masking Description: The assessor and statistician will be blinded to randomisation outcomes and will perform assessments on all participants from both arms. Assessments will be conducted at two time points: at the completion of the program (UCIR or RITH) and at six weeks following initial hospital admission. This blinding minimises potential bias in outcome evaluation and ensures the integrity, reliability, and objectivity of the trial's findings.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation in the Home (RITH) (Experimental): Participants randomised to the experimental pathway. Participants will receive home-based therapy from a multidisciplinary (MDT) team, including physiotherapists, occupational therapists, social workers, dieticians, medical practitioners, psychologists, and pharmacists.
  Interventions: Other: Rehabilitation in the home
- Usual Care Inpatient Rehabilitation (UCIR) (Active Comparator): Participants randomised to the usual care pathway. Participants will receive care in a rehabilitation ward or subacute hospital, including therapy from a multidisciplinary team.
  Interventions: Other: Usual care inpatient rehabilitation

INTERVENTIONS:
Other: Rehabilitation in the home — Participants will receive home-based therapy from a MDT team, including physiotherapists, occupational therapists, social workers, dietitians, medical practitioners, psychologists, and pharmacists. Participants will be transferred to RITH once they achieve a level of mobility (+/- assistance) that enables them to manage at home. As per usual care, the disciplines required, frequency of visits, duration of visits, and duration of rehabilitation will be based on the patient's specific needs. There will be weekly MDT conferences to discuss patient progress led by medical staff. Telehealth care may be incorporated into the RITH program, subject to patient preference and provider availability. If the participant deteriorates during the RITH program, the escalation plan mandated by the LHD HITH Department will be followed to ensure appropriate care is provided. As for UCIR, discharge occurs when patients achieve sufficient walking and functional ability with available assistance.
  Arms: Rehabilitation in the Home (RITH)
Other: Usual care inpatient rehabilitation — Participants will receive care in a rehabilitation ward or subacute hospital, including therapy from a MDT team. Discharge occurs when patients achieve sufficient walking and functional ability with available assistance, typically within 1-3 weeks, though this varies.
  Arms: Usual Care Inpatient Rehabilitation (UCIR)

SUMMARY:
Hip fractures are common, especially in older adults, and they can have a big impact on health and quality of life. In Australia, hip fractures are a significant healthcare challenge. After surgery, patients often need rehabilitation to regain mobility, but this usually involves long hospital stays. The RITH4Hips trial will determine if a program where patients receive rehabilitation at home (instead of in the hospital) is similar to conventional inpatient rehabilitation.

Objectives:

The main goal of this study is to find out if rehabilitation at home after surgery for a hip fracture works as well as rehabilitation in the hospital. The investigators also want to see if the home rehabilitation program can reduce the time spent in a hospital bed and improve other aspects like quality of life, mobility, and pain management.

Methods:

This study will involve older adults who have had surgery due to a low-trauma hip fracture. Participants will be randomly assigned to either the usual care inpatient rehabilitation or the Rehabilitation in the Home (RITH) program. The investigators will measure outcomes such as how well patients can move, how much pain they experience, how their quality of life improves, and how much time they spend in the hospital.

Expected Outcomes:

The investigators expect that the home rehabilitation program will be just similar to inpatient rehabilitation in helping patients recover mobility. The investigators also hope to find that it will reduce the time patients spend in a hospital bed, improve their quality of life, reduce fear of falling, and lessen the burden on carers. Additionally, the investigators aim to show that the home program is more cost-effective than hospital-based rehabilitation.

DETAILED DESCRIPTION:
Study Aim This study aims to determine whether a multidisciplinary Rehabilitation in the Home (RITH) program for patients following low-trauma hip fracture (LTHF) is non-inferior to inpatient rehabilitation in terms of mobility during activities of daily living (ADL), assessed using the de Morton Mobility Index (DEMMI)

Study Design This is a pragmatic, multicentre, randomised, single-blinded, parallel-group, non-inferiority clinical trial with an embedded qualitative component.

As part of recruitment monitoring, reasons for declining participation will be recorded for individuals approached but not enrolled.

Hypotheses

The investigators hypothesise that compared to inpatient rehabilitation, the RITH program will be:

Non-inferior in terms of mobility recovery (DEMMI score within 2.9 points). Superior in reducing hospital bed days, with at least a 6-day reduction in physical ward stay.

Superior in improving health-related quality of life, walking ability, fear of falling, opioid consumption, and carer experience.

More cost-effective than usual care. Effective in reducing total length of stay (LOS), provided barriers to rapid transition to RITH are addressed.

Methods

Eligibility is determined perioperatively.

Inclusion criteria

* Adults aged ≥50 admitted to Liverpool or Bankstown hospitals with LTHF who:
* Undergo surgical management.
* Were living in the community pre-injury and plan to return home.
* Weight bear as tolerated post-surgery.
* Are deemed suitable for rehabilitation.
* The presence of a carer, if required for mobility or function, is necessary at the time of transfer to the community. The carer must be prepared to manage the patient within 3 days post-randomisation.
* Suitable environment for home-based rehabilitation as assessed by the MDT as per usual practice.

Once cleared for rehabilitation (typically 5-10 days post-surgery), participants will be randomised to:

Intervention Groups

Usual Care Inpatient Rehabilitation (UCIR): Participants will receive care in a rehabilitation ward or subacute hospital, including therapy from a multidisciplinary team. Discharge occurs when they achieve sufficient walking and functional ability, typically within 1-3 weeks. Researchers will collect information about carer visits and associated costs during the stay.

Rehabilitation in the Home (RITH): Participants will receive therapy at home from a multidisciplinary team. Discharge occurs when they achieve sufficient walking and functional ability, typically within 1-3 weeks. Researchers will contact patients about carer-related costs during the program.

Follow-up Assessments:

After completing rehabilitation, researchers will visit participants at home (or in the clinic if preferred) shortly after discharge and again six weeks after their initial hospital admission to assess walking ability, daily activities, confidence, quality of life, pain, and post-surgery challenges. Researchers will also gather information on healthcare visits, costs, and new community services used. If participants have carers, the carers will be invited to complete a voluntary survey about carer experience. Medical records will also be reviewed to understand the care provided over the study period.

Qualitative study:

A purposive sample of patients and their carers who were randomised to the RITH group will be invited to participate in a one-on-one interview some weeks after completing rehabilitation. Additionally, an opportunistic sample of other stakeholders such as clinicians, healthcare managers, and insurers will be invited to participate. The embedded qualitative study seeks to gain insights into why the RITH program was or was not deemed effective for individual participants, as well as how the RITH program may be made more acceptable for future implementation.

Sample size calculation:

A sample of 220 participants (allowing for 7% loss to follow-up) is required to detect:

A 2.9-point between-group difference in DEMMI (non-inferiority margin: 6, SD: 8.9).

A 6-day reduction in hospital bed days (mean 25, SD 17, negative binomial parameter theta = 2.1) with 80% power (α = 0.05).

Analysis plan for primary outcome: The primary outcome will be analysed using an analysis of covariance (ANCOVA) with the 6-week DEMMI score as the dependent variable, and independent variables of group, timepoint, and an interaction between group and timepoint. The 6-week DEMMI will be examined using contrasts of the interaction.

Cost analysis: A cost-effectiveness analysis will be conducted alongside this trial, including both direct and indirect costs.

Analysis plan for qualitative study: Qualitative interviews will be analysed using the Rapid Assessment Process, combining deductive and inductive approaches for efficient thematic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adults ages ≥ 50 years presenting to Liverpool hospital or Bankstown-Lidcombe hospital with a low-trauma (osteoporotic) hip fracture who undergo surgical management
* Anticipated to return to community (private) residence
* Permitted to weight-bear as tolerated post-surgery
* Suitable for inpatient rehabilitation (i.e., requires multidisciplinary rehabilitation, is considered cognitively suitable by the MDT to participate in the rehabilitation program being examined, and would otherwise be admitted to inpatient rehabilitation)
* The presence of a carer, if required for mobility or function, is necessary at the time of transfer to the community. The carer must be prepared to manage the patient within 3 days post-randomisation. This time frame is considered necessary as carers will not be able to complete all required preparations before randomisation, and allowing an extended preparation period could bias the length of physical ward bed stay for the RITH group
* Suitable environment for home-based rehabilitation as assessed by the MDT as per usual practice

Exclusion Criteria:

* Presence of a concomitant condition that precludes actively participating in a rehabilitation program at home
* Residential location outside the Bankstown-Canterbury, Liverpool, and Fairfield Local Government Areas
* Active end-of-life management or palliative care
* Previously participated in the HITH4Hips or RITH4Hips trials

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-09-20 (Estimated)

PRIMARY OUTCOMES:
De Morton Mobility Index (DEMMI) | At 1 to 3 days following discharge from the rehabilitation program (an average of 14 days after admission to rehabilitation) and at 6 weeks after initial admission.
  The De Morton Mobility Index is a mobility outcome measure specifically designed for an older population. The DEMMI assesses 15 tasks which are associated with activities of daily living such as bed mobility and sit-to-stand transitions. The DEMMI is scored between 0 - 100, where 0 represents no mobility and 100 represents full mobility. The Minimal Clinically Important Difference (MCID) for the DEMMI is estimated to be approximately 6 points, representing the smallest change necessary to reflect a clinically meaningful improvement in mobility.

SECONDARY OUTCOMES:
Length of Stay (LOS) - Total | At 1 to 3 days following discharge from the rehabilitation program (an average of 14 days after admission to rehabilitation).
  Number of days spent in the program, from acute admission until discharge from rehabilitation.
Length of Stay (LOS) - Physical Ward Bed | At 1 to 3 days following discharge from the rehabilitation program (an average of 14 days after admission to rehabilitation).
  Number of days spent in a physical ward bed in the hospital (including both acute and subacute locations).
Index Hip Pain | Assessments will occur at baseline (within 24 hours prior to randomisation), daily during the allocated rehabilitation program (an average of 14 days from admission to rehabilitation), and at 6 weeks following initial hospital admission.
  Hip pain at rest, on movement, and maximum. Score is a numerical rating from 0 - 10, where 0 is no pain and 10 is the worst pain imaginable.
EuroQol-5D-5L (EQ5D) | Assessments will be conducted at baseline (within 24 hours prior to randomisation), at 1 to 3 days following discharge from the rehabilitation program (an average of 14 days after admission to rehabilitation), and at 6 weeks post-admission.
  The EuroQol-5D-5L is a questionnaire used to measure patient's health-related quality of life. It assesses 5 domains related to mobility, self-care, usual activities, pain/discomfort and anxiety/depression and provides a score between 1 - 5 for each domain where 1 means no problems, and 5 means extreme problems.
Timed Up-and-Go Test (TUG Test) | At 1 to 3 days following discharge from the rehabilitation program (an average of 14 days after admission to rehabilitation) and at 6 weeks after initial admission.
  The Timed Up-and-Go Test measures the time required for a patient to stand from a seated position and walk three meters at a comfortable pace using any required mobility aids, before returning to a seated position. The TUG Test is a good indicator of overall mobility and fall risk, however, it will only be used on patients deemed capable of safely conducting this test.
Falls Efficacy Scale (FES) | At 1 to 3 days following discharge from the rehabilitation program (an average of 14 days after admission to rehabilitation) and at 6 weeks after initial admission.
  The Falls Efficacy Scale is a 10-item questionnaire used to assess a patient's fear of falling during various activities of daily living. Each item is scored between 1 - 10, where 1 means very confident with this activity, and 10 means not confident at all with this activity. Higher scores indicate a higher fear of falling.
Zarit Carer Burden Interview (ZCBI) | At 1 to 3 days following discharge from the rehabilitation program (an average of 14 days after admission to rehabilitation).
  The short-form Zarit Carer Burden Interview assesses the physical, emotional, social, and financial burden associated with being a caregiver. Each item is assigned a score from 0 - 4, where 0 means never and 4 means nearly always. Higher total scores are associated with increased carer burden.
Positive Aspects of Caregiving Scale (PACS) | At 1 to 3 days following discharge from the rehabilitation program (an average of 14 days after admission to rehabilitation).
  The Positive Aspects of Caregiving Scale assesses the perceived benefits experienced by caregivers as a result of their role. The PACS is designed to balance to conventionally negatively-skewed burden assessments by instead focusing on domains related to personal growth and relationship satisfaction. The PACS uses a scale of 1 - 5 for each item where 1 means strongly disagree and 5 means strongly agree. Higher total scores are associated with more positive caregiving experiences.
Functional Independence Measure (FIM) | At 1 to 3 days following discharge from the rehabilitation program (an average of 14 days after admission to rehabilitation) and at 6 weeks after initial admission.
  The Functional Independence Measure (FIM) is a routinely used outcome measure in inpatient rehabilitation to assess a patient's level of disability and need for assistance with activities of daily living. It consists of 18 items, each scored on a 1-7 scale, where 1 indicates total assistance required and 7 signifies complete independence. Higher total scores reflect greater overall functional independence.
Hospital-Acquired Complications (HACs) | At 1 to 3 days following discharge from the rehabilitation program (an average of 14 days after admission to rehabilitation).
  The rate and types of Hospital-Acquired Complications (HACs) will be recorded at the end of the program, with definitions aligned to the Australian Commission on Safety and Quality in Health Care (https://www.safetyandquality.gov.au/our-work/indicators-measurement-and-reporting/hospital-acquired-complications-hacs). Additionally, regular safety monitoring of adverse events will be conducted throughout the program.

OTHER OUTCOMES:
Quality-Adjusted Life Years (QALYs) | Assessments will be calculated at 6 weeks post-admission.
  QALYs will be derived from responses to the EQ-5D questionnaire administered at three timepoints: baseline (prior to randomisation), 1 to 3 days after discharge from the rehabilitation program, and 6 weeks post-admission. This measure will quantify patient health outcomes and quality of life over time, enabling the evaluation of the RITH program's impact on patient well-being.
Health Service Costs | Health service costs will be assessed using data from each hospital's Finance Department, covering admission to the end of the allocated rehabilitation program (average 14 days post-rehab admission). Data will be available 8 to 12 weeks post-discharge.
  The total episode of care cost to the health service will be assessed from the provider's perspective. Episode of care costs will be obtained directly from the hospital, while direct costs for each episode of care and episode of service will be sourced from the health service. All costs will be adjusted to 2025 values using the Gross Domestic Price Index.
Participant and Carer Costs | Assessments will occur weekly during the allocated rehabilitation program (up to average 14 days from rehabilitation admission), and at 6 weeks following initial hospital admission.
  Participant and carer costs will be collected through regular follow-ups and will include expenses such as costs for parking, transportation, home modifications, medication, and lost productivity due to time taken off work. These costs will capture the financial burden on both participants and their carers as part of the economic evaluation of the RITH program.
Incremental Cost-Effectiveness Ratio (ICER) | Assessments will be calculated at 6 weeks following initial hospital admission.
  The ICER will be calculated as the cost per additional Quality-Adjusted Life Year (QALY) gained, comparing the health service cost and participant and carer costs of the RITH and UCIR programs. This measure will assess the cost-effectiveness of the RITH program by evaluating the economic impact relative to improvements in patient health outcomes.
Opioid Consumption | Assessments will occur daily through completion of the allocated rehabilitation program, starting on Day 1 and continuing until discharge (on an average duration of 14 days), and at 6 weeks following initial hospital admission.
  Opioid consumption throughout the program duration will be recorded in oral morphine equivalent daily dose (OMEDD), using the opioid calculator developed by the Faculty of Pain Medicine, Australian and New Zealand College of Anaesthetists. Additionally, opioid use at 6 weeks post-admission will be measured as a yes/no outcome. For participants reporting continued opioid use at 6 weeks, the frequency and reason for use will also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Thuy Anh Bui, BSC, GradCert Higher Ed, PhD, Principal Investigator — South West Sydney Local Health District
Locations (3):
- Australia (3):
  - Liverpool Hospital, Sydney, New South Wales
  - Fairfield Hospital, Sydney, New South Wales
  - Bankstown-Lidcombe Hospital, Sydney, New South Wales

IPD SHARING:
Plan to Share IPD: Yes
De-identified Individual Participant Data (IPD) will be shared in accordance with the ICMJE policy. The study protocol will be shared as a publication. Specifically, de-identified data from this study will be securely stored in a REDCap database, accessible only to authorised researchers with approval from the South West Local Health District Human Research Ethics Committee. Paper-based records will be securely maintained, and no identifying information will be disclosed in any publications or reports, ensuring full compliance with privacy and ethical standards. Upon reasonable request, de-identified data from this study may be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: De-identified Individual Participant Data (IPD) for this study will be available for sharing within 15 years after the study closure. Qualitative data will be securely stored for 5 years from the date of any publication, during which it will be available for sharing. After this period, the data will be destroyed in a confidential manner.
Access Criteria: Access to Individual Participant Data (IPD) will be granted to authorised researchers who meet the following criteria:
  Researchers must provide a scientific rationale for requesting data, including the type of analysis to be conducted, with statistical methods subject to independent review approval.
  A data sharing proposal must be submitted, outlining the planned analyses and data required.
  A data sharing agreement must be signed, specifying the terms of use and confidentiality.
  Proposals and agreements will be submitted via email. Access will only be granted once these conditions are met.